CLINICAL TRIAL: NCT03483987
Title: Re-treatment of Chronic Hepatitis C Virus Infection Among Non-responders or Those Who Relapsed to Treatment With Regimens Based on Direct-acting Antiviral Drugs
Brief Title: Re-treatment of HCV Following DAA Failure
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in recruiting the participants
Sponsor: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government)
Collaborators: Ram Manohar Lohia Institute of Medical Sciences, Lucknow (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-202-IP-100
Record Dates: First submitted 2018-03-24; First posted 2018-03-30 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2021-04

CONDITIONS: Chronic Hepatitis C
Keywords: Hepatitis c virus; Direct acting antiviral drugs; Virological relapse
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C

STUDY DESIGN:
Intervention Model Description: Participants who relapsed to prior treatment with one or two DAA will be retreated with second course of DAA regimen and ribavirin with or without pegylated interferon. The duration of treatment will be 24 weeks. The drugs will be chosen based upon their prior exposure to DAA, liver disease severity and virus genotype.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sof+Ledi+R arm (Experimental): Participants with HCV genotype 1,4, 5 or 6 and relapsed with following regimens will be treated with sofosbuvir, ledipasvir and ribavirin combination
  1. Sofosbuvir plus velpatasvir with or without ribavirin for 12 weeks
  2. Sofosbuvir plus ribavirin with or without pegylated interferon for 12 or 24 weeks
  3. Sofosbuvir plus velpatasvir with or without ribavirin for 24 weeks and are not eligible for pegylated interferon
  Interventions: Drug: Sof+Ledi+R arm
- Sof+Ledi+R+Peg-IFN arm (Experimental): Participants with HCV genotype 1,4, 5 or 6, who have relapsed after a 24 weeks treatment regimen of sofosbuvir plus velpatasvir with or without ribavirin combination and are eligible for pegylated interferon, will be treated with a combination of sofosbuvir, ledipasvir, ribavirin plus pegylated interferon
  Interventions: Drug: Sof+Ledi+R+Peg-IFN arm
- Sof+Dacla+R arm (Experimental): Participants with HCV genotype 2 or 3 and relapsed with following regimens will be treated with a combination of sofosbuvir, daclatasvir and ribavirin
  1. Sofosbuvir plus velpatasvir with or without ribavirin for 12 weeks
  2. Sofosbuvir plus ribavirin with or without pegylated interferon for 12 or 24 weeks
  3. Sofosbuvir plus velpatasvir with or without ribavirin for 24 weeks and are not eligible for pegylated interferon
  Interventions: Drug: Sof+Dacla+R arm
- Sof+Dacla+R+Peg-IFN arm (Experimental): Participants with HCV genotype 2 or 3, who have relapsed after a 24 weeks treatment regimen of sofosbuvir plus velpatasvir with or without ribavirin combination and are eligible for pegylated interferon, will be treated with a combination of sofosbuvir, ledipasvir, ribavirin plus pegylated interferon
  Interventions: Drug: Sof+Dacla+R+Peg-IFN arm
- Sof+Velpa+R arm (Experimental): Following group of participants will be treated with sofosbuvir, velpatasvir and ribavirin combination
  1. who were treated earlier with 12 week treatment regimen of either sofosbuvir plus daclatasvir or sofosbuvir plus ledipasvir with or without ribavirin or
  2. who were earlier treated with a 24 treatment regimen of either sofosbuvir plus daclatasvir or sofosbuvir plus ledipasvir with or without ribavirin and are not eligible for pegylated interferon
  Interventions: Drug: Sof+Velpa+R arm
- Sof+Velpa+R+Peg-IFN arm (Experimental): Participants, who have relapsed after a 24 week treatment regimen of either sofosbuvir plus daclatasvir or sofosbuvir plus ledipasvir with or without ribavirin and are eligible for pegylated interferon will be treated with sofosbuvir, velpatasvir, ribavirin and pegylated interferon combination
  Interventions: Drug: Sof+Velpa+R+Peg-IFN arm

INTERVENTIONS:
Drug: Sof+Ledi+R arm — Fixed dose combination of sofosbuvir 400 mg plus ledipasvir 90 mg once daily plus ribavirin 1000 mg (body weight <75 kg) or 1200 mg (body weight =>75 kg) daily in two divided doses
  Other Names: SLR
  Arms: Sof+Ledi+R arm
Drug: Sof+Ledi+R+Peg-IFN arm — Fixed dose combination of sofosbuvir 400 mg plus ledipasvir 90 mg once daily plus ribavirin 1000 mg (body weight <75 kg) or 1200 mg (body weight =>75 kg) daily in two divided doses plus pegylated interferon alpha 2b @ 1.5 microgram/kg subcutaneously once in a week
  Other Names: SLR+Peg
  Arms: Sof+Ledi+R+Peg-IFN arm
Drug: Sof+Dacla+R arm — Sofosbuvir 400 mg once daily plus daclatasvir 100 mg once daily plus ribavirin 1000 mg (body weight <75 kg) or 1200 mg (body weight =>75 kg) daily in two divided doses
  Other Names: SDR
  Arms: Sof+Dacla+R arm
Drug: Sof+Dacla+R+Peg-IFN arm — Sofosbuvir 400 mg once daily plus daclatasvir 100 mg once daily plus ribavirin 1000 mg (body weight <75 kg) or 1200 mg (body weight =>75 kg) daily in two divided doses plus pegylated interferon alpha 2b @ 1.5 microgram/kg subcutaneously once in a week
  Other Names: SDR+Peg
  Arms: Sof+Dacla+R+Peg-IFN arm
Drug: Sof+Velpa+R arm — Fixed dose combination of sofosbuvir 400 mg plus velpatasvir 100 mg once daily plus ribavirin 1000 mg (body weight <75 kg) or 1200 mg (body weight =>75 kg) daily in two divided doses
  Other Names: SVR
  Arms: Sof+Velpa+R arm
Drug: Sof+Velpa+R+Peg-IFN arm — Fixed dose combination of sofosbuvir 400 mg plus velpatasvir 100 mg once daily plus ribavirin 1000 mg (body weight <75 kg) or 1200 mg (body weight =>75 kg) daily in two divided doses plus pegylated interferon alpha 2b @ 1.5 microgram/kg subcutaneously once in a week
  Other Names: SVR+Peg
  Arms: Sof+Velpa+R+Peg-IFN arm

SUMMARY:
HCV infection is treated with oral drugs, termed as 'direct-acting anti-viral agents' (DAAs). In India, four DAAs are available (sofosbuvir [SOF], daclatasvir [DCV], ledipasvir [LDV] and velpatasvir [VEL]). Globally, DAA based regimens have obtained excellent rates of cure. Cure of HCV infection is defined as undetectable HCV RNA 12 weeks after stopping drugs, also referred to as sustained virological response at week 12 (SVR12).

Using these DAA based treatment regimens, a small number (up to 5%) of people fail to achieve SVR12 and HCV RNA reappear after a few weeks of stopping the drugs (virological relapse). Data on management of virological relapse are extremely limited, especially in genotype 3, and no guidelines exist regarding re-treatment options for such group. Hence, we plan to re-treat such people using what appear to be the best combination treatment in each situation and to review our experience over time.

Participants with chronic HCV infection who relapsed following standard DAA-based treatment regimen will be invited to participate. We propose to re-treat them with the anti-HCV drug combination which appears to be the most suited to his/her clinical profile, based on the current empiric knowledge - the choice of drugs will be based on HCV genotype, the previous treatment regimen and the presence/absence of liver cirrhosis, etc.

During anti-HCV treatment, participants will be given expected standard of care and HCV RNA will be tested at 4-week intervals starting from week 4 and till RNA becomes undetectable, and then at the end of treatment and 12 weeks after the treatment was stopped - as is the usual practice during such treatment. Relevant clinical, laboratory and treatment details will be recorded in a pre-defined data collection form. Treatment outcome will be categorized as success (SVR12), treatment failure (any detectable HCV RNA at the end of 24 weeks treatment duration) or relapse (HCV RNA negative at the end of treatment, but positive at 12 weeks after stopping treatment).

If possible, a 5-ml blood specimen will be collected before starting re-treatment from all participants; in addition, another similar specimen will be collected following the treatment in those in whom the re-treatment is unsuccessful. These will be stored and may be used in future for virological studies to look for drug-resistance variations.

DETAILED DESCRIPTION:
-Introduction Oral drugs, termed collectively as 'Direct-acting anti-viral agents' (DAAs), are the standard-of-care for HCV treatment. In India, four DAAs, namely sofosbuvir (SOF), daclatasvir (DCV), ledipasvir (LDV) and velpatasvir (VEL), are marketed. Initially, people were treated using SOF in combination with ribavirin with or without pegylated-interferon (Peg-IFN). Thereafter, HCV treatment was switched to use of two DAAs with or without ribavirin and discontinuation of Peg-IFN. All these combinations of DAAs have obtained excellent rates of cure - defined as undetectable HCV RNA at 12 weeks after stopping DAA-based HCV, also referred to as sustained virological response at week 12 (SVR12).

Though DAAs-based anti-HCV treatment has shown generally excellent results, globally some patients fail to achieve SVR12. The rate of such failure is higher in patients with advanced liver disease and HCV genotype 3 infections. In India, genotype 3 is the most prevalent HCV genotype (~65%), followed by genotype 1 (~30%).

Data on management of the people who relapse after DAA treatment are extremely limited, and no guidelines exist regarding retreatment options for them. Hence, physician need to re-treat such people with the best combination available in a given situation.

* Objective To study the re-treatment response in people with chronic HCV infection and relapsed to prior DAA based treatment
* Rationale for the proposed treatment regimens

Overall, investigators attempted to tried to combine drugs to give the best chance of virus clearance to those with prior treatment failure by following the following principles, as have emerged from the experience worldwide:

1. Prolongation of treatment duration to 24 weeks if previous treatment was for 12 weeks
2. Addition of pegylated interferon (previous standard of care for HCV, and which acts by a different mechanism) if person has previously failed 24 weeks of dual-DAA treatment
3. Addition of ribavirin, if it appears that the participant can tolerate this drug.
4. Use of sofosbuvir (a NS5b inhibitor) as the backbone of re-treatment, since drug resistance to this drug is the least common
5. Use of a pangenotypic drug (velpatasvir) if the previous treatment was with a genotype-specific NS5a inhibitor (daclatasvir or ledipasvir)
6. Use of genotype-specific drug (daclatasvir or ledipasvir) if the previous treatment was with a pan-genotypic NS5a inhibitor (velpatasvir)

   * Methods Relevant clinical, laboratory and treatment details will be recorded in pre-defined data collection form, used for monitoring patients with HCV infection as part of their clinical care. Treatment outcome will be categorized as successful (SVR12), treatment failure (any detectable HCV RNA at the end of pre-defined 12-24 weeks treatment duration) or relapse (HCV RNA negative at the end of treatment, but positive at 12 weeks after stopping treatment). The data will be analyzed for the entire group and for specific subgroups, such as: (i) those without cirrhosis; (ii) those with compensated cirrhosis; (iii) those with decompensated cirrhosis
   * Blood specimen collection If possible, a 5 ml blood specimen will be collected before starting anti-HCV retreatment from all the participants. If the HCV retreatment also fails, then a repeat 5 ml blood specimen will be collected for virological studies.
   * Follow-up plan During anti-HCV treatment: HCV RNA will be tested at 4-week intervals starting from week 4 till RNA reports are negative, and then at the end of treatment and 12 weeks after stopping treatment.
   * Sample size Considering usual clinical load, investigators expect to treat around 1000-1200 DAA treatment naive people with chronic HCV infection between during the study period. considering a 5% relapse rate, HCV relapse is expected in about 50 people.

ELIGIBILITY:
Inclusion Criteria:

* participants with chronic HCV infection and viremia, who have completed the DAA-based standard treatment and relapsed
* regardless of severity of liver disease, HCV genotype, nature or duration of DAAs,and whether treatment-naïve or previously treated with Peg-IFN/ribavirin

Exclusion Criteria:

1. Participants with chronic kidney disease
2. Post-organ transplant recipients
3. Short life expectancy (<1 year)
4. Not willing to follow-up
5. Individuals with immunocompromised states: HIV, immunosuppressive drugs, cancer chemotherapy, congenital hemolytic anemia

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-02-10 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
SVR12 | - 12 weeks after stopping 24 weeks of DAA based treatment
  Proportion of participants with undetectable HCV RNA at 12 weeks after stopping DAA-based HCV re-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Aggarwal, DM, Principal Investigator — Sanjay Gandhi Postgraduate Institute of Medical Sciences (SGPGI)
Locations (2):
- India (2):
  - Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow, Uttar Pradesh
  - RML Institute of Medical Sciences, Lucknow, Uttar Pradesh

IPD SHARING:
Plan to Share IPD: No
Presently, we have no plan to share data with other researchers

REFERENCES:
- [Derived] Goel A, Katiyar H, Mayank, Tiwari P, Rungta S, Verma A, Deep A, Sana A, Rai P, Aggarwal R. Hepatitis C Retreatment With First-Line Direct Acting Antiviral Drugs. J Clin Exp Hepatol. 2023 Sep-Oct;13(5):736-741. doi: 10.1016/j.jceh.2023.03.007. Epub 2023 Mar 24. PMID 37693269